CLINICAL TRIAL: NCT00952770
Title: Effect of Statins on the Progression of the Intima-media Thickness of the Radial Artery After Radial Angioplasty
Brief Title: Effect of Statins on the Radial Intima-media Thickness After Transradial Angioplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chungnam National University (Other)
Responsible Party: Jae-Hyeong Park, MD, PhD, Chungnam National University, Chungnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CNUH-09-07-60
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Coronary intervention; intima-media thickness
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Experimental): Group receiving atorvastatin 20mg/day
  Interventions: Procedure: transradial coronary intervention
- Simvastatin/Ezetimibe (Active Comparator): Group receiving simvastatin/ezetimibe 10/10mg
  Interventions: Procedure: transradial coronary intervention

INTERVENTIONS:
Procedure: transradial coronary intervention — percutaneous coronary intervention with transradial approach

SUMMARY:
The first event of the atherosclerotic plaque formation is the accumulation of the low density lipoprotein-cholesterol (LDL-cholesterol) in to the intima of the arterial wall. After accumulation of the LDL-cholesterol, the oxidation of the LDL-cholesterol particles and recruitment of monocytes to the intima and media are the next steps. The thickening of intima-media thickness (IMT) is resulted from these initial events. The IMT can be easily measured by high-resolution ultrasonography in various arteries including carotid, brachial and radial arteries. The increased carotid IMT can be used as a non-invasive independent parameter indicating increased cardiovascular mortality. Some investigators reported increased radial IMT is associated with increased early failure of the radiocephalic arteriovenous fistula in the hemodialysis patients. Moreover, radial IMT is increased in patients underwent radial artery intervention because of denudation injury of the radial artery. Recently, the use of statin can halt the progression of the carotid IMT progression. However, it is unknown that the use of statin can prevent the progression of radial IMT after the transradial coronary intervention. The investigators want to evaluate the effect of statins on the progression of the radial IMT after the transradial intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary intervention via the radial artery

Exclusion Criteria:

* Contraindication to statins
* Left ventricular ejection fraction less than 30%
* Recent history of hematologic disease or leukocyte count <3000/mm3 and/or platelet <100 000/mm3
* Hepatic dysfunction with AST or ALT >3 times the upper normal reference limit
* History of renal dysfunction or a serum creatinine level >2.0 mg/dL
* Serious noncardiac comorbid disease with a life expectancy <1 year
* Inability to follow the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Difference of IMT between two groups | 1 month, 6 months

SECONDARY OUTCOMES:
Difference of epicardial fat thickness Difference of cholesterol level | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Hyeong Park, MD, PhD, Principal Investigator — Chungnam National University, Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea